CLINICAL TRIAL: NCT01934998
Title: Characterization of the Parkinsonism and Other Non-ataxia Spectrum and Striatal Dopaminergic Degeneration in Spinocerebellar Ataxia Type 6
Brief Title: Parkinsonism in Spinocerebellar Ataxia Type 6
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 12-1335
Record Dates: First submitted 2013-08-27; First posted 2013-09-04 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Spinocerebellar Ataxia Type 6
Keywords: SCA6, parkinsonism, Datscan
MeSH Terms: conditions — Spinocerebellar Ataxias; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SCA6 and control: SCA6 and control
- SCA6 or controls: Twelve SCA6 patients and 8 controls to be studied

SUMMARY:
The spinocerebellar ataxias (SCAs) are a genetically heterogeneous group of dominantly inherited progressive ataxia disorders. More than 30 different gene loci have been identified so far. The most common SCAs, which together account for more than half of all affected families, are SCA1, SCA2, SCA3, and SCA6. Each of these disorders is caused by a translated CAG repeat expansion mutation. SCA1, SCA2, and SCA3 usually have an onset between 30 and 40, and SCA6 usually begins at the age of 50 to 60. In addition to progressive ataxia, SCA1, SCA2, and SCA3 frequently present with additional non-ataxic symptoms, including parkinsonism. Carbidopa/levodopa was found to have a good therapeutic effect on parkinsonism.

The SCA6 used to be considered a pure cerebellar disorder. However, a recent large study on natural history of SCAs found that patients with SCA6 often had nonataxia symptoms, an observation that challenges the view that SCA6 is a purely cerebellar disorder. Parkinsonism in SCA6 was rarely reported, except in a case serial, or a small size study in Korean patients.

Dopamine transporter (DAT) is a very reliable dopaminergic neuronal marker. Reduction in DAT density detected by I123 SPECT DaTscanTM in the dopaminergic neuron terminal striatum was reported in one small size study consisting of eight SCA6 patients in Korea. There was also a PET study using different radioligand for DAT in a small group of SCA6 patients in Germany, which found sub-clinical change in DAT density in some patients with SCA6.

There has been no study so far in the US on parkinsonism and other non-ataxia spectrum and striatal dopaminergic damage in SCA6, probably because non-ataxia feature of SCA6 hasn't received much attention, and also because DaTscanTM hasn't been clinically available in US until recently. The only two published studies on SCA6 and DAT were from Korea and Germany, which were of small subject size. There has been no treatment available for SCA6 so far.

Our hypothesis is that parkinsonism and other non-ataxia spectrum and striatal dopaminergic neurodegeneration are part of the SCA6 disease spectrum.

DETAILED DESCRIPTION:
Specifically, we would expect to see

1. Parkinsonism and other non-ataxia symptoms are more commonly present in SCA6 patients than we used to think.
2. Parkinsonism is associated with the loss of DAT in striatum.
3. Parkinsonism and other non-ataxia symptoms are also associated with the expanded allele repeat number, the disease duration, and the severity of ataxia, in addition to DAT loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older with progressive ataxia and positive genetic test for SCA6 will be recruited. Those who take medications known to affect DAT binding, such as Ritalin, Cocaine, and Adderall will be excluded. Those taking SSRIs for depression will be asked to stop the medications for at least 24 hours before the DaTscanTM. All study patients will have the decision making capability to understand the study and requirements and consent for themselves.

The age-matched controls will most likely be the patients' spouses. However friends or family members may also serve as controls if needed. Control subjects will have no ataxia, parkinsonism, myoclonus and other focal neurological symptoms and deficits.

Exclusion Criteria:

* Subjects who don't meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SCA6 patients and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome would be the clinical feature of the parkinsonism and change in DAT density in putamen and caudate | 10 months
  The UPDRS-II and -III scores

SECONDARY OUTCOMES:
The secondary outcome would be the INAS score | 10 months
  INAS score and its association with the DAT density and UPDRS scores
The secondary outcome would also be the SARA score | 10 months
  The SARA score and its association with the DAT density and UPDRS scores

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xie, MD PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States